CLINICAL TRIAL: NCT02198703
Title: RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED CLINICAL TRIAL FOR EVALUATING THE EFFICACY OF AB-LIFE PROBIOTIC PRODUCT ON THE LDL-CHOLESTEROL REDUCTION IN THE MODERATE HYPERCHOLESTEROLEMIA
Brief Title: A Trial to Evaluate the Efficacy of AB-Life Probiotic Product on LDL-Cholesterol Reduction in Moderate Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AB-Life study #3
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2015-09

CONDITIONS: Moderate Hypercholesterolemia
Keywords: Probiotics; AB-Life; LDL-cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AB-Life (Experimental): 1 capsule of AB-Life daily during 12 weeks consumed immediately before, after or during the breakfast. The daily dose corresponds to the intake of 1.8E+10 CFU. According to the product's stability and the duration of the experiment, all participants receive at least 1.2E+09 CFU/capsule/day by the end of the study.
  Interventions: Dietary Supplement: Probiotics bacterial strains
- Placebo (Placebo Comparator): 1 capsule of placebo daily during 12 weeks consumed immediately before, after or during the breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics bacterial strains
  Other Names: AB-Life
  Arms: AB-Life
Dietary Supplement: Placebo
  Other Names: AB-life
  Arms: Placebo

SUMMARY:
This study aims to demonstrate the effect of the chronic consumption of AB-Life probiotic blend on blood LDL cholesterol level in volunteers with moderate hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to the study, male and female volunteers will have to fulfill the following criteria (assessment based on the medical examination performed at V1 with a checking at V3):

* Age between 18 and 65 years (limits included).
* BMI between 18,5 and 30 kg/m² ((limits excluded).
* For women : Non menopausal with reliable contraception since at least two cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom alone without spermicide gel and oestrogenic contraceptive excluded) or menopausal without oestrogenic replacement therapy.
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination.
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form.
* Affiliated with a social security scheme.
* Agree to be registered on the volunteers in biomedical research file.

After V1 biological analysis the subjects will be eligible to the visit V2 on the following criteria:

- Fasting plasma LDLc level (Friedewald estimation method) between 1,3 and 1,89 g/L (3,35 - 4,92 mmol/L, limits included with ± 2% tolerated around).

After V2 biological analysis the subjects will be eligible to the study on the following criteria:

- Fasting plasma LDLc level (Friedewald estimation method) between 1,3 and 1,89 g/L (3,35 - 4,92 mmol/L, limits included with ± 2% tolerated around).

A re-screening can occur from 2 months after the exit of study for failure to comply with the one or more of the eligibility criteria listed above.

Exclusion Criteria:

Volunteers with the following criteria will be considered as non eligible to the study (assessment based on the medical examination performed at V1 with a checking at V3):

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other chronic severe disease.
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease).
* With a history of ischemic cardiovascular event or, during the previous 6 months a surgical procedure.
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient.
* Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg).
* Pregnant or lactating women or intending to become pregnant within 5 months ahead.
* Under lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 4 months before the randomization.
* Under medication which could affect blood lipid parameters (e.g. long-term corticosteroid systemic drug, systemic antibodies, androgens or phenytoin, etc.) or stopped less than 1 month before the randomization (stable long-term treatment with beta blocker or thiazide diuretics tolerated).
* Regular intake of dietary supplements or "functional foods" which may interfere with lipid absorption and/or metabolism (e.g. rich in plant stanol or sterol like PRO-ACTIV or DANACOL products, red yeast rice, policosanol, omega-3 fatty acids like fish oils, ST HUBERT OMEGA 3 or PRIMEVERE products, soya protein, oat fiber like QUAKER OATS, psyllium, chitosan, guar gum, inulin, etc.) or stopped less than 3 months before the randomization.
* Under treatment which could disturb microbiota balance or stopped in a too short period before the randomization (e.g. less than one month for laxatives, less than 6 weeks for antibiotics).
* Regular intake of dietary supplements or "functional foods" containing prebiotics, probiotics or symbiotics (e.g. BION 3, LACTIBIANE, ACTIMEL, ACTIVIA, etc.) or stopped less than 1 month before the randomization.
* Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the randomization.
* With significant change in food habits or in physical activity in the 3 months before randomization or not agreeing to keep them unchanged throughout the study.
* With reported body weight variation > 5% in the 3 months prior the randomization or with a hyper or hypocaloric diet planned in the next 5 months.
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator.
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 standard drinks daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study.
* Smoking more than 10 cigarettes daily or not agreeing to keep his smoking habits unchanged throughout the study.
* Recent history of chronic alcohol or drug abuse (in the last 2 years).
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded).
* Who made a blood donation in the 3 months before the randomization or intending to make it within 4 months ahead.
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial.
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros.
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision.
* Presenting a psychological or linguistic incapability to sign the informed consent.
* Impossible to contact in case of emergency.

After V1 biological analysis the subjects will be considered as non eligible to the study on the following criteria :

* Fasting plasma glucose level > 1,26 g/L (6,99 mmol/L).
* Fasting plasma triglycerides > 3,5 g/L (3,95 mmol/L).
* Fasting plasma TC, HDLc or insulin with an abnormality judged as clinically significant according to the investigator.

After V2 biological analysis the subjects will be considered as non eligible to the study on the following criteria:

* Fasting plasma TC, HDL or TG with an abnormality judged as clinically significant according to the investigator.
* Serum AST, ALT, GGT, ALP or bilirubin with an abnormality judged as clinically significant according to the investigator.
* Serum urea or creatinine with an abnormality judged as clinically significant according to the investigator.
* Complete blood count with clinically significant abnormality according to the investigator.

Volunteers with the following criteria at the V3 will be considered as non eligible to the study:

* Capsules' consumption less than 80% of capsules during the run-in period (since V1) according to the quantities returned.
* Gastroenteritis history finished less than 2 weeks before the randomization.

The included subjects who cannot be randomized at V3 because of a too short wash out period related to the non inclusion criteria E8, E10, E12 or E34 can delay their visit V3 without to exceed 28 days from the visit V2.

A re-screening can occur from 2 months after the exit of study for failure to comply with the one or more of the eligibility criteria listed above (except for E33 criteria).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of the fasting blood LDL cholesterol concentration | 12 weeks

SECONDARY OUTCOMES:
Change in fasting blood total cholesterol concentration | 4 weeks
Change in fasting blood total cholesterol concentration | 12 weeks
Change in fasting blood LDLc concentration | 4 weeks
Change in fasting blood HDLc concentration | 4 weeks
Change in fasting blood HDLc concentration | 12 weeks
Change in fasting blood ratio total cholesterol / HDLc concentrations | 4 weeks
Change in fasting blood ratio total cholesterol / HDLc concentrations | 12 weeks
Change in fasting blood ratio LDLc / HDLc concentrations | 4 weeks
Change in fasting blood ratio LDLc / HDLc concentrations | 12 weeks
Change in fasting blood triglycerides concentration | 4 weeks
Change in fasting blood triglycerides concentration | 12 weeks
Change in fasting blood Apo A1 concentration | 4 weeks
Change in fasting blood Apo A1 concentration | 12 weeks
Change in fasting blood Apo B100 concentration | 4 weeks
Change in fasting blood Apo B100 concentration | 12 weeks
Change in fasting blood insulin concentration | 4 weeks
Change in fasting blood insulin concentration | 12 weeks
Change in fasting blood glucose concentration | 12 weeks
Change in fasting blood glucose concentration | 4 weeks
Change in fasting blood acetate concentration | 12 weeks
Change in fasting blood propionate concentration | 12 weeks
Change in fasting blood acetate / propionate concentrations | 12 weeks
Change in SCORE - European Low Risk Chart of fatal cardiovascular disease | 4 weeks
Change in SCORE - European Low Risk Chart of fatal cardiovascular disease | 12 weeks
Change in fasting blood hsCRP concentration | 12 weeks
Complete blood count | 12 weeks
Blood Alkaline Phosphatase | 12 weeks
Blood Alanine Amino Transferase | 12 weeks
Blood Aspartate Amino Transferase | 12 weeks
Blood Gamma Glutamyl Transpeptidase | 12 weeks
Blood total bilirubin | 12 weeks
Blood urea | 12 weeks
Blood creatinine | 12 weeks
Heart rate | 4 weeks
Heart rate | 12 weeks
Systolic Blood Pressure | 4 weeks
Diastolic Blood Pressure | 4 weeks
Diastolic Blood Pressure | 12 weeks
Systolic Blood Pressure | 12 weeks
Body weight | 4 weeks
Body weight | 12 weeks
Physical Activity Score | 12 weeks
Total energy intake | 12 weeks
Percentage of energy intake from fat | 12 weeks
Dietary fiber intake | 12 weeks
Saturated Fatty Acids intake | 12 weeks

OTHER OUTCOMES:
Fasting blood PCSK9 concentration | 12 weeks
Fasting blood FGF-19 concentration | 12 weeks
Fasting blood LDLox concentration | 12 weeks
Fasting blood fibrinogen concentration | 12 weeks
Fasting blood biliary acids concentrations | 12 weeks
Fecal concentrations of neutral sterol including cholesterol and its secondary metabolites | 12 weeks
Fecal concentrations of phytosterols | 12 weeks
Fecal concentrations of volatil fatty acids | 12 weeks
Fecal concentrations of branched chain fatty acids | 12 weeks
Fecal concentrations of biliary acids | 12 weeks
Fecal concentrations of AB-Life probiotic strains | 12 weeks
Fecal concentration of calprotectin | 12 weeks
Fasting blood sodium concentration | 12 weeks
Fasting blood potassium concentration | 12 weeks
Fasting blood bicarbonates concentration | 12 weeks
Fasting blood calcium concentration | 12 weeks
Fasting blood inorganic phosphate concentration | 12 weeks
Urine aspect | 12 weeks
Urine color | 12 weeks
Urinary density level | 12 weeks
Urinary bilirubin level | 12 weeks
Urinary urobilirubinogen level | 12 weeks
Urinary protein level | 12 weeks
Urinary glucose level | 12 weeks
Urinary ketones level | 12 weeks
Urinary nitrites level | 12 weeks
Urine sediment | 12 weeks
Urine osmolality | 12 weeks
Urine pH | 12 weeks
Urinary red cells level | 12 weeks
Urinary white cells level | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Gendre, M.D., Principal Investigator — BioFortis; Ariana Salavert, Ph. D., Study Director — AB-BIOTICS
Locations (2):
- France (2):
  - Naturalpha, Lille
  - Biofortis, Saint-Herblain